CLINICAL TRIAL: NCT02090920
Title: Individualized Dosing of Nifedipine for Tocolysis in Preterm Labor
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Sara Quinney, Sara Quinney, Pharm D, PhD, Indiana University
Other Study IDs: 1106006106
Record Dates: First submitted 2014-03-03; First posted 2014-03-18 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Nifedipine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma for determination of nifedipine and oxidized nifedipine concentrations Blood for DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nifedipine: Nifedipine 10 mg immediate release tablet by mouth loading dose Nifedipine administered orally every 15-20 minutes for the first hour to a maximum loading dose of 30 mg, followed by a maintenance dose of 10-20 mg immediate release nifedipine administered orally every 6 hours
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Nifedipine — Nifedipine 10 mg immediate release tablet by mouth loading dose Nifedipine administered orally every 15-20 minutes for the first hour to a maximum loading dose of 30 mg, followed by a maintenance dose of 10-20 mg immediate release nifedipine administered orally every 6 hours
  Other Names: Adalat, Nifediac, Nifedical, Procardia, Procardia XL

SUMMARY:
This study looks at the effects of a mother's genes and other characteristics (mother's age, baby's age, race, and other diseases) on the ability of nifedipine to end contractions and prevent an early delivery. This information will be used to decide what amount of nifedipine women need to best treat preterm contractions.

DETAILED DESCRIPTION:
The purpose of this study is to identify the relationship between the amount of nifedipine in a woman's body and its effect on ending preterm (early) labor contractions and delaying delivery by at least 48 hours. The study will also look at the effects of genes (materials passed from parent to child that determine the make-up of the body) and other characteristics (for example mother's age, baby's age, race, and other diseases or drugs) on the ability of nifedipine to end the contractions. We will use this information to decide what amount of nifedipine women need to best treat preterm contractions. This study will also examine the effect of pregnancy on how fast nifedipine is removed from the woman's body.

This study will be conducted on two phases. The first will study women who are starting nifedipine for treatment of preterm labor. Nifedipine dose will be determined by the patient's physician. Blood samples will be obtained from the mother to determine the concentration of nifedipine and its metabolite, oxidized nifedipine, during one dosing interval. A blood sample will also be obtained for DNA isolation to examine variants in genes involved in the nifedipine pathway. We will also collect data on uterine contractions and blood pressure through clinical monitoring. After delivery, maternal and umbilical cord blood samples will be obtained, along with a piece of placenta. Women who take part in the first phase will be asked to return 6-10 weeks after delivery. At that time, she will take a single dose of 10 mg immediate release nifedipine by mouth and blood samples will be collected for up to 6 hours. Blood pressure will also be monitored prior to collection of each blood sample

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years of age or older
* Diagnosed with preterm labor (defined as 1-3 uterine contractions per 10 minute interval for at least 60 minutes with evidence of change in cervical dilation and/or effacement)
* Prescribed nifedipine as a tocolytic agent
* Signed informed consent

Exclusion Criteria:

* Multifetal gestation
* Cervical dilation of 5 cm or greater
* Ruptured uterine membranes
* Any medical or obstetrical condition that would contraindicate tocolytic therapy including placental abruption; placenta previa; nonreassuring fetal status; uterine growth restriction; severe congenital abnormalities
* Administration of medications known to interact with CYP3A (a human gene) other than betamethasone or dexamethasone as indicated for stimulating fetal lung maturation, within the past 24 hours unless approved by study investigators
* Administered a potent mechanism-based CYP3A inhibitor (e.g. erythromycin, clarithromycin) in past 48 hours
* History of allergy or hypersensitivity to nifedipine
* History of taking grapefruit or grapefruit juice by mouth within the last 24 hours
* Known current hepatic or renal disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant Women with preterm labor who have been prescribed immediate release nifedipine and admitted at Eskenazi Health Hospital or Indiana University Methodist Hospital.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
prevention of delivery for 48 hours with attainment of uterine quiescence | One Year
  The primary study outcome is prevention of delivery for 48 hours with attainment of uterine quiescence, defined by 12 hours of six or fewer contractions per hour and no further cervical change. Failure of the primary outcome occurs if, in the first 48 hours, patients deliver, rupture membranes, experience recurrent preterm labor, continue to contract or experience cervical change, or required the use of alternate tocolytics. Secondary outcomes include time to uterine quiescence (≤6 contractions/hour), birth weight, gestational age at delivery, maternal and neonatal adverse effects.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Quinney, PharmD, PhD, Principal Investigator — Indiana University Clinical Pharmacology
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - IU Health Methodist, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided